CLINICAL TRIAL: NCT01010477
Title: Double-Blind, Placebo-Controlled Trial of Nicotine Nasal Spray as an Aid for Smoking Cessation in Schizophrenia
Brief Title: Trial of Nicotine Nasal Spray as an Aid for Smoking Cessation in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01DA024640-01A1 (NIH); 1R01DA024640-01A1 (NIH)
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Smoking Cessation; Schizophrenia
Keywords: smoking cessation; schizophrenia; nicotine nasal spray; behavioral counseling
MeSH Terms: conditions — Smoking Cessation; Schizophrenia | interventions — Tobacco Use Cessation Devices; Nicotine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine Nasal Spray (Experimental): Subjects will be instructed to use the nasal spray at a minimum of 8 doses each day and up to a maximum of 5 doses per hour and 40 doses in 24 hours starting on the TQD. Subjects will be instructed to use the nasal spray at a minimum of 8 doses each day and up to a maximum of 5 doses per hour and 40 doses in 24 hours starting on the TQD. . Nasal spray will be used from the TQD through the end of Week 20.
  Interventions: Drug: Nicotine Nasal Spray; Behavioral: Behavioral counseling
- Placebo nasal spray (Placebo Comparator): Subjects will be instructed to use the nasal spray at a minimum of 8 doses each day and up to a maximum of 5 doses per hour and 40 doses in 24 hours starting on the TQD. Subjects will be instructed to use the nasal spray at a minimum of 8 doses each day and up to a maximum of 5 doses per hour and 40 doses in 24 hours starting on the TQD. Nasal spray will be used from the TQD through the end of Week 20.
  Interventions: Drug: Nicotine Nasal Spray; Behavioral: Behavioral counseling

INTERVENTIONS:
Drug: Nicotine Nasal Spray — minimum 8 doses of nasal spray per day; maximum of 5 doses per hour, no more than 40 doses per day
  Other Names: Nicotrol
Behavioral: Behavioral counseling — Both groups will receive behavioral intervention designed for schizophrenia delivered as 15 individual counseling sessions over 26 weeks.

SUMMARY:
This R01 grant describes a randomized, double-blind, placebo-controlled trial of nicotine nasal spray (NNS) as an aid for smoking cessation in 60 individuals with schizophrenia. The objectives of this study are to determine the efficacy of NNS with behavioral intervention for smoking cessation in smokers with schizophrenia. It is hypothesized that the quit rate of subjects who receive NNS and behavioral intervention will be significantly greater than the quit rate of the control group who will receive the placebo spray plus same behavioral intervention. Quit rate is defined as the proportion of individuals who self report no tobacco use during weeks 5 through 8 confirmed by exhaled carbon monoxide (CO) less than 10 parts per million during these 4 weeks. The investigators will also assess abstinence rates at Study Weeks 12 and 20 on the NNS and at weeks 26 and 52 after the medication has been stopped. Since studies of this group suggest high relapse rates when treatments are discontinued (Evins et al., 2005; George et al., 2000; George et al., 2002a), the investigators will continue NNS treatment for a total of 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be invited to participate in the study if they fulfill the following inclusion criteria:

  1. Meet DSM-IV diagnostic criteria for Schizophrenia
  2. Be 18 years of age or older
  3. Be daily smokers of 10 or more cigarettes per day (cpd)
  4. Have an expired CO level > 9 ppm
  5. Be motivated to quit smoking
  6. Be willing to adhere to the study protocol (e.g. provide samples, attend all visits)
  7. Be able to give informed consent
  8. Stable on their current atypical antipsychotic medication for at least one month.

Exclusion Criteria:

* Subjects will be excluded based on any one of the following exclusion criteria:

  1. Current suicidal risk, including active suicidal ideation, recent suicidal behavior or suicide attempt in the past 30 days,
  2. Psychiatric hospitalization in the last 30 days
  3. Inability to read or understand the questionnaires in English
  4. Current pregnancy or lactation or plans to become pregnant in the next 12 months
  5. Regular use of non-cigarette forms of tobacco including cigars, pipes, smokeless tobacco
  6. Patients with significant cognitive impairment that may interfere with their study participation assessed as a Folstein Mini-Mental Status exam score of less than 22.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Williams, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 141 subjects screened. Of these 66 were consented. Eleven were later found to be ineligible and were dropped prior to randomization. Fifty five subjects were randomized to active or placebo NNS. Three subjects were found to be not eligible after randomization leaving 52 for analysis.
Groups:
- NNS Active: Receives active nicotine containing Nasal spray
- Placebo: Receives placebo (piperine)nasal spray
Period: Overall Study
Arm/Group | NNS Active | Placebo
Started | 27 | 25
Completed | 21 | 22
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- NNS Active: Receives nicotine (active) nasal spray
- Placebo NS: Receives placebo (piperine containing) nasal spray
- Total: Total of all reporting groups
Arm/Group | NNS Active | Placebo NS | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.8) | 48.4 (10.5) | 45.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 18 | 14 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 13 | 27
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Quit Smoking From Weeks 5 to 8
Description: Quit rate is defined as the proportion of individuals who self report no tobacco use during weeks 5 through 8 confirmed by exhaled carbon monoxide (CO) less than 10 parts per million (ppm) during these 4 weeks.
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- NNS Active: Receives nicotine (active ) nasal spray
Arm/Group | NNS Active | Placebo
Number analyzed (Participants) | 27 | 25
participants | 3 | 1
Statistical Analysis 1: Comparison: NNS Active vs Placebo; Fisher Exact test (2-sided); Test type: Superiority or Other; p = 0.632, Fisher Exact — threshold for statistical significance: p< 0.05

ADVERSE EVENTS:
Time Frame: adverse event data were collected for 1 year
Arm/Group | NNS Active | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 18/27 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NNS Active (N=27) | Placebo (N=25)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 18 | 6
throat irritation (Ear and labyrinth disorders) | 12 | 1

LIMITATIONS AND CAVEATS:
small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No